CLINICAL TRIAL: NCT00983034
Title: Prospective Study of the Effects of Helicobacter Pylori Eradication on Renal Functions and Proteinuria in Patients With Membranous Nephropathy
Brief Title: The Effects of Helicobacter Pylori Eradication on Proteinuria in Patients With Membranous Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Yasar Caliskan, Division of Nephrology, Department of Intenal Medicine, Istanbul Faculty of Medicine, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20061976
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Nephrotic Syndrome; Glomerulonephritis; Membranous Nephropathy
Keywords: nephrotic syndrome; Helicobacter pylori infection; proteinuria; membranous nephropathy
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulonephritis; Glomerulonephritis, Membranous; Proteinuria | interventions — Lansoprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Membranous nephropathy (Active Comparator): Patients with primary membranous nephropathy diagnosed by biopsy
  Interventions: Drug: lansoprazole, amoxicillin, clarithromycin
- IgA nephropathy (Active Comparator): Patients with IgA nephropathy diagnosed by biopsy
  Interventions: Drug: lansoprazole, amoxicillin, clarithromycin
- Focal segmental glomerulosclerosis (Active Comparator): Patients with primary focal segmental glomerulosclerosis diagnosed by biopsy
  Interventions: Drug: lansoprazole, amoxicillin, clarithromycin

INTERVENTIONS:
Drug: lansoprazole, amoxicillin, clarithromycin — lansoprazole, 30 mg twice daily, plus amoxicillin, 0.75 g twice daily, plus clarithromycin, 250 mg twice daily, for 14 days

SUMMARY:
Membranous nephropathy (MN) may also be secondary to many other diseases (e.g., infections, drugs, neoplasms and autoimmune diseases). In this study, the presence of Helicobacter Pylori (H. pylori) antigen was investigated in renal tissue from needle biopsy samples, and the prevalence of H. pylori infection and the effects of H. pylori eradication on proteinuria level in patients with MN will be investigated.

DETAILED DESCRIPTION:
Membranous nephropathy (MN) is a common cause of nephrotic syndrome in adults. It is thought to be mainly a primary or idiopathic form; however, it may also be secondary to many other diseases (e.g., infections, drugs, neoplasms and autoimmune diseases). In this study, the presence of Helicobacter Pylori antigen was investigated in renal tissue from needle biopsy samples, and the prevalence of H. pylori infection and the effects of H. pylori eradication on proteinuria level in patients with MN will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Nondiabetic patients
* Patients with primary glomerulonephritis
* Clinical diagnosis of membranous nephropathy, IgA nephropathy or focal segmental glomerulosclerosis confirmed by biopsy
* Glomerular filtration rate > 30 mL/min
* Patients who did not receive Helicobacter pylori eradication therapy within the last three months before enrollment in study

Exclusion Criteria:

* Patients with secondary glomerulonephritis
* Glomerular filtration rate < 30 mL/min
* Patients who received Helicobacter pylori eradication therapy within the last three months before enrollment in study
* Patients with a history of gastric surgery
* Patients without an informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Daily proteinuria levels after Helicobacter Pylori eradication treatment | 6 months

SECONDARY OUTCOMES:
Glomerular filtration rate | 6 months
Serum creatinine level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, MD, Principal Investigator — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University; Berna Yelken, MD, Principal Investigator — Division of Nephrology, Istanbul Faculty of Medicine, Istanbul University; Halil Yazici, MD, Principal Investigator — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University; Mehmet S Sever, Prof MD, Study Director — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University
Locations (1):
- Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Caliskan B, Yazici H, Caliskan Y, Ozluk Y, Gulluoglu M, Kilicaslan I, Turkmen A, Sever MS. The Effects of Helicobacter pylori Eradication on Proteinuria in Patients with Primary Glomerulonephritis. Int J Nephrol. 2014;2014:180690. doi: 10.1155/2014/180690. Epub 2014 Feb 24. PMID 24707402